CLINICAL TRIAL: NCT01063231
Title: Evaluation of PillCam™ Colon 2 in Visualization of the Colon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MA-201
Record Dates: First submitted 2009-10-18; First posted 2010-02-05 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2010-11

CONDITIONS: Colonic Diseases; and Large Bowel Diseases
Keywords: Colonic Diseases; bowel diseases
MeSH Terms: conditions — Colonic Diseases; Intestinal Diseases | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Subjects that are indicated for colonoscopy, who are suspected or known to suffer from large bowel diseases.
  Interventions: Device: PillCam™ (Capsule Endoscopy) Colon 2 capsule

INTERVENTIONS:
Device: PillCam™ (Capsule Endoscopy) Colon 2 capsule — Medical Device

SUMMARY:
Evaluate accuracy of PCCE-2 in detecting patients with colonic polyps as compared to conventional colonoscopy.

DETAILED DESCRIPTION:
Standard evaluation of subjects with suspected colon diseases includes endoscopic imaging by colonoscopy and radiology testing such as: air-contrast barium enema, abdominal/pelvic CT, or virtual colonoscopy.

The Given® Diagnostic System offers an alternative approach for endoscopic visualization of the colon. Advantages of the Given® Diagnostic System include the elimination of the need for conscious sedation, the minimally invasive, painless nature of the exam, and the ability to pursue normal daily activities immediately following the procedure . Furthermore, compared to standard colonoscopy, the Given® Diagnostic System may be more readily accepted by the subjects, thereby improving subjects' willingness to undergo a diagnostic evaluation of the colon and comply with colorectal cancer screening recommendations.

The PillCam™ SB capsule (formerly M2A® Capsule) that was cleared by the FDA- in August 2001 for small bowel evaluation has been ingested to date by more than 1,000,000 people worldwide and is well accepted by patients and physicians as well as the professional societies. However, adequate visualization of the colon cannot be achieved with the standard PillCam™ SB capsule because of the anatomical and physiological properties of the colon which are significantly different than the small bowel. Moreover, other issues that limit the evaluation of the colonic mucosa by the standard PillCam™ SB procedure include an unsatisfactory level of colon cleanliness and slow progression of the PillCam™ SB capsule through the colon during the desired examination time. Therefore, the development and introduction of a specially designed, customized colon capsule combined with a dedicated capsule colonoscopy procedure protocol will allow for more efficient evaluation of the colonic mucosa. This is expected to improve the capability of the Given® Diagnostic System to detect colonic pathologies and to serve as a diagnostic and screening tool for colonic disease. To date, several clinical studies have been conducted with Given® Diagnostic System and the PillCam™ Colon 1 capsule A pilot multicenter study is currently being conducted with a new Given® Diagnostic System and an advanced generation of the the PillCam™ Colon capsule - PillCam™ Colon 2. Capsule. The new development of Given® Diagnostic System and PillCam™ Colon 2 capsule is primarily aimed to increase sensitivity and specificity for polyp detection.

Further details of the Given® Diagnostic System and PillCam™ Colon 2 capsule can be found in the device description section.

This study is designed to evaluate the performance of the new version of Given® Diagnostic System and PillCam™ Colon 2 capsule in detecting patients with polyps and other colonic lesions as compared to conventional colonoscopy.

ELIGIBILITY:
Inclusion criteria:

* Subject is between the ages of 18-80
* Subject was referred to colonoscopy for at least one of the following reasons:

  * Colorectal cancer screening for age ≥50
  * Clinical symptoms such as: rectal bleeding, hematochezia, melena, positive FOBT, recent change of bowel habits for age ≥50
  * Positive findings in the colon (e.g. Polyp ≥10mm)
  * Personal history of polyps that were removed at least 3 years ago (3 years and above)

Exclusion criteria

* Subject has dysphagia or any swallowing disorder
* Subject has congestive heart failure
* Subject has high risk of renal insufficiency associated with the use of sodium phosphate
* Subject is not eligible for colon preparation due to the presence of underlying conditions based on the clinical judgment of the investigator
* Subject has any allergy or other known contraindication to the medications used in the study
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
* Subject has a cardiac pacemaker or other implanted electro medical device.
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject with any condition believed to have an increased risk for capsule retention such as Crohn's disease, intestinal tumors, radiation enteritis, incomplete colonoscopies due to obstructions or NSAID enteropathy,
* Subject with gastrointestinal motility disorders
* Subject has known delayed gastric emptying
* Subject has any condition, which precludes compliance with study and/or device instructions.
* Women who are either pregnant at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
* Subject suffers from life threatening conditions
* Subject currently participating in another clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Accuracy parameters of PillCam™ COLON 2 in detecting patients with colonic polyps ≥6mm and ≥10 mm as compared to conventional colonoscopy | within 7 days

SECONDARY OUTCOMES:
Diagnostic yield of PillCam™ COLON 2 in detecting colonic lesions as compared to conventional colonoscopy | within 7 days
Assessment of colon cleansing level at different colon segments for PillCam and Colonoscopy | within 7 days
Distribution of capsule excretion time up to 10 hours post ingestion based on Rapid videos | within 7 days
Capsule transit time within stomach, small bowel and colon based on Rapid videos | within 7 days
Prevalence of polyps at different size categories and locations as detected by capsule and by conventional colonoscopy | Within 7 days
RAPID reading time Number, type and severity of adverse events | with in 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Guido Costamagna, Prof., Principal Investigator — Ospedale Gemelli; Guido Costamagna, Prof, Principal Investigator — Ospedale Gemelli
Locations (8):
- Hospital Erasme - Gastro-Enterologie, Brussels, Belgium
- France (2):
  - Chef de Service dHepato-Gastro-Enterologie et dAssistance Nutritionnelle CHU Nantes, Nantes
  - CHU Nancy, Vandœuvre-lès-Nancy
- Evangelisches Krankenhaus, Düsseldorf, Germany
- Ospedale Gemelli,ENDOSCOPIA DIGESTIVA, Roma, Italy
- Academic Medical Center University of Amsterdam, Amsterdam, Netherlands
- Clinica Universitaria de Navarra, Pamplona, Spain
- Malmo University Hospital, Malmo, Sweden